CLINICAL TRIAL: NCT02591836
Title: An 8-Week, Double-Blind, Randomized, Placebo-Controlled, Dose-Ranging Study of the Efficacy and Safety of Gemcabene Administered as Monotherapy or in Combination With Atorvastatin in the Treatment of Hypercholesterolemic Patients
Brief Title: Efficacy and Safety of Gemcabene in Hypercholesterolemic Patients as Monotherapy or in Combination With Atorvastatin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NeuroBo Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A4141001
Record Dates: First submitted 2015-10-22; First posted 2015-10-30 (Estimated); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Hypercholesterolemia
Keywords: LDL-C; Lipid Regulator
MeSH Terms: conditions — Hypercholesterolemia | interventions — gemcabene; Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (16):
- Gemcabene 300 mg (Experimental): Gemcabene 300 mg QD
  Interventions: Drug: Gemcabene
- Gemcabene 600 mg (Experimental): Gemcabene 600 mg QD
  Interventions: Drug: Gemcabene
- Gemcabene 900 mg (Experimental): Gemcabene 900 mg QD
  Interventions: Drug: Gemcabene
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Atorvastatin 10 mg (Active Comparator)
  Interventions: Drug: Atorvastatin
- Atorvastatin 40 mg (Active Comparator)
  Interventions: Drug: Atorvastatin
- Atorvastatin 80 mg (Active Comparator)
  Interventions: Drug: Atorvastatin
- Gemcabene 300 mg & Atorvastatin 10 mg (Experimental)
  Interventions: Drug: Gemcabene; Drug: Atorvastatin
- Gemcabene 300 mg & Atorvastatin 40 mg (Experimental)
  Interventions: Drug: Gemcabene; Drug: Atorvastatin
- Gemcabene 300 mg & Atorvastatin 80 mg (Experimental)
  Interventions: Drug: Gemcabene; Drug: Atorvastatin
- Gemcabene 600 mg & Atorvastatin 10 mg (Experimental)
  Interventions: Drug: Gemcabene; Drug: Atorvastatin
- Gemcabene 600 mg & Atorvastatin 40 mg (Experimental)
  Interventions: Drug: Gemcabene; Drug: Atorvastatin
- Gemcabene 600 mg & Atorvastatin 80 mg (Experimental)
  Interventions: Drug: Gemcabene; Drug: Atorvastatin
- Gemcabene 900 mg & Atorvastatin 10 mg (Experimental)
  Interventions: Drug: Gemcabene; Drug: Atorvastatin
- Gemcabene 900 mg & Atorvastatin 40 mg (Experimental)
  Interventions: Drug: Gemcabene; Drug: Atorvastatin
- Gemcabene 900 mg & Atorvastatin 80 mg (Experimental)
  Interventions: Drug: Gemcabene; Drug: Atorvastatin

INTERVENTIONS:
Drug: Gemcabene — Gemcabene
  Arms: Gemcabene 300 mg; Gemcabene 300 mg & Atorvastatin 10 mg; Gemcabene 300 mg & Atorvastatin 40 mg; Gemcabene 300 mg & Atorvastatin 80 mg; Gemcabene 600 mg; Gemcabene 600 mg & Atorvastatin 10 mg; Gemcabene 600 mg & Atorvastatin 40 mg; Gemcabene 600 mg & Atorvastatin 80 mg; Gemcabene 900 mg; Gemcabene 900 mg & Atorvastatin 10 mg; Gemcabene 900 mg & Atorvastatin 40 mg; Gemcabene 900 mg & Atorvastatin 80 mg
Drug: Atorvastatin — Atorvastatin
  Arms: Atorvastatin 10 mg; Atorvastatin 40 mg; Atorvastatin 80 mg; Gemcabene 300 mg & Atorvastatin 10 mg; Gemcabene 300 mg & Atorvastatin 40 mg; Gemcabene 300 mg & Atorvastatin 80 mg; Gemcabene 600 mg & Atorvastatin 10 mg; Gemcabene 600 mg & Atorvastatin 40 mg; Gemcabene 600 mg & Atorvastatin 80 mg; Gemcabene 900 mg & Atorvastatin 10 mg; Gemcabene 900 mg & Atorvastatin 40 mg; Gemcabene 900 mg & Atorvastatin 80 mg
Drug: Placebo
  Arms: Placebo

SUMMARY:
The primary purpose of this placebo-controlled study is to evaluate the low-density lipoprotein cholesterol (LDL-C) efficacy and dose-response of gemcabene 300, 600 and 900 mg/day administered as monotherapy or in combination with atorvastatin 10, 40, and 80 mg/day to hypercholesterolemic patients.

Secondary purposes include evaluating the effects of high-sensitivity C-reactive protein (hsCRP), high-density lipoprotein cholesterol (HDL-C), triglycerides (TG) and apolipoprotein B (ApoB), and safety and efficacy of gemcabene monotherapy and gemcabene/atorvastatin combination.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females
* 18-70 years old
* Received a statin as monotherapy while having a LDL-C >100 mg d/L at initial clinical washout visit OR
* Received no lipid-altering drugs since the initial clinic washout visit and had a mean LDL-C as follows at 2 qualifying visits:
* ≥ 130 mg/dL if National Cholesterol Education Program (NCEP) Adult Treatment Panel III (ATP III) Coronary Heard Disease (CHD) risk ≥ 10%; OR
* ≥ 160 mg/dL if NCEP ATP III CHD risk < 10%
* Had variability of 2 qualifying LDL-C <20% (i.e. lowest value/highest value >0.8). An additional qualifying visit may have been completed by patients who were washing off lipid medication in order to reassess LDL-C variability; and
* Had a mean LDL-C < 250 mg/dL at 2 qualifying visits

Exclusion Criteria:

* Women of childbearing potential, pregnant or lactating;
* Body Mass Index (BMI) >38kg/m²;
* TG >400 mg/dL at Visit B2 or B3
* Unexplained creatinine phosphokinase (CPK) > 3 x Upper Limit of Normal (ULN) or those with a history of unexplained myopathy (including rhabdomyolysis);
* Documented cardiac history of: Myocardial infarction*, severe or unstable angina pectoris, coronary angioplasty, coronary artery bypass graft, symptomatic carotid artery disease or peripheral artery disease, ventricular arrhythmias, recurrent supraventricular tachycardia, abnormal QTC interval (QT corrected > 0.44 sec), heart failure or any other major cardiovascular event resulting in hospitalization
* Uncontrolled hypertension*
* Type 1 diabetes mellitus or uncontrolled type 2 diabetes mellitus (HbA1c >8%) or any diabetic patient who takes insulin and/or thiazolidinediones
* Renal dysfunction including chronic renal failure or insufficiency, or creatinine >2.0 mg/dL;
* Hepatic dysfunction
* Uncontrolled hypothyroidism
* Abnormal urinalysis
* Currently taking any of the following medications:
* Potent CYP3A4 inhibitors including indinavir, nelfinavir, ritonavir, saquinavir, amiodarone, cimetidine, clarithromycin, erythromycin, erythromycin, fluoxetine, itraconazole, ketoconazole, nefazodone and troleandomycin as well as grapefruit juice;
* Thiazolidinediones (Avandia, Actos);
* Immunosuppressive agents;
* St. John's wort
* Taking any of the following lipid-altering medications within 5 weeks prior to randomization:
* Lipid-regulating drugs: Niacin (crystalline >500mg/day, slow release or time release), psyllium preparation such as Metamucil (>2 tablespoons/day), fibrates and derivatives, bile cholesterol absorption inhibitors including ezetimibe;
* Any supplement containing plan sterols/stanols (i.e. Benecol, beta-sitosterol, Cholestatin, Phytoquest, Take Control) or cholestin (i.e. Chinese red yeast, fermented on rice; Hong Qu, Hong Chu, Herbvalin, Ruby Monascus, Monascus purpureus rice);
* Neomycin (oral);
* Adrenocortical steroids*
* Sibutramine (Meridia);
* Insulin;
* Orlistat (Xenical);
* Isotretinoin

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 277 (Actual)
Dates: Start 2003-01; Primary Completion 2003-06 (Actual); Study Completion 2003-06 (Actual)

PRIMARY OUTCOMES:
LDL-C percent change from baseline | 56 days

SECONDARY OUTCOMES:
HDL-C percent change from baseline | 56 days
TG percent change from baseline | 56 days
Apolipoprotein-B percent change from baseline | 56 days
Adverse Events | 56 days
Clinical Laboratory | 56 days
  Clinical Laboratory Abnormalities